CLINICAL TRIAL: NCT02500095
Title: Substrate Metabolism, Growth Hormone Signaling, and Insulin Sensitivity During Fasting in Overweight and Obese Human Subjects and the Impact of Growth Hormone Receptor Blockade
Brief Title: Substrate Metabolism, Growth Hormone Signaling, and Insulin Sensitivity During Fasting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: fasting8000
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — Angptl4 protein, mouse; Sodium Chloride; pegvisomant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): 12 hours of fasting
- Fasting and saline (Experimental): 72 hours of fasting and concomitant saline
  Interventions: Other: Fasting; Drug: Saline
- Fasting and GHR blockade (Experimental): 72 hours of fasting and concomitant Growth hormone receptor (GHR) blockade with Pegvisomant (Somavert) for inhibition of the fasting-induced GH secretion
  Interventions: Other: Fasting; Drug: Pegvisomant

INTERVENTIONS:
Other: Fasting — 72 hours of fasting
  Arms: Fasting and GHR blockade; Fasting and saline
Drug: Saline — Concomitant saline during fasting
  Arms: Fasting and saline
Drug: Pegvisomant — Concomitant Growth hormone receptor blockade with Pegvisomant during fasting
  Arms: Fasting and GHR blockade

SUMMARY:
Background: Calorie restriction increases longevity in many species and attenuate the development of chronic disorders including type 2 diabetes, cardiovascular diseases and cancer. In mice reduced activity of insulin-like growth factor I (IGF-I) and/or insulin is associated with extended longevity. Growth hormone (GH) is the main regulator of IGF-I production, but the molecular mechanism whereby GH switches from IGF-I stimulation (protein anabolism) to fatty acid oxidation (fatty acid catabolism) as well as induction of insulin resistance during fasting remains enigmatic.

Hypotheses: The changes of the global set of metabolites, induction of insulin resistance, and the shift in metabolism from protein anabolism to lipolysis together with the potentially favorable effect of calorie restriction during fasting depend on preserved fasting-induced GH secretion.

Aim: The investigators wish to provide knowledge on changes in metabolites and shift in signaling pathways that take place at the transition to the fasting state among healthy overweight and obese subjects. Furthermore the investigators wish to determine the effect of GH on the adaption of the metabolism to a fasting state.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* written consent
* body mass index (BMI) 25-40
* age 20-60 years

Exclusion Criteria:

* any kind of disease
* regular medication

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Insulin and growth hormone signaling, expressed as CHANGE in phosphorylation of intracellular target proteins and CHANGE in messenger ribonucleic acid (mRNA) expression of target genes in muscle- and fat-tissue. | Muscle and fat biopsies obtained at t1= 9.00 am (60 min) and t2=12.30 am (270 min) on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days)
  Change in phosphorylation of target proteins and mRNA expression of target genes

SECONDARY OUTCOMES:
Glucose metabolism | Change in glucose metabolism using glucose tracer from t=0 min - 360 min on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days)
  Change in glucose metabolism assessed by tracer kinetics on every study day and by indirect calorimetry.
Magnetic resonance (MR) spectroscopy | During fasting: t= 12 hours and t= 48 hours of fasting
Change in concentrations of metabolites in the insulin and growth hormone signaling pathways using metabolomics | Muscle-tissue obtained at t1= 9.00 am (60 min) and t2=12.30 am (270min) on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days)
  Method: Metabolomics
Fat metabolism | Change in fat metabolism using palmitic acid tracer from t1=180 min - 240 min and t2=300 min - 360 min on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days)
  Change in fat metabolism assessed by tracer kinetics on every study day and by indirect calorimetry.
Protein metabolism | Change in protein metabolism using urea tracer from t=0 min - 240 min on each study day after 0, 4 and 8 weeks (interval of 4 weeks between each of the three study days)
  Change in protein metabolism assessed by tracer kinetics on every study day and by indirect calorimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor, Principal Investigator — Aarhus University / Aarhus University Hospital; Jens Otto L. Jørgensen, Professor, Study Chair — Aarhus University / Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Hogild ML, Gudiksen A, Pilegaard H, Stodkilde-Jorgensen H, Pedersen SB, Moller N, Jorgensen JOL, Jessen N. Redundancy in regulation of lipid accumulation in skeletal muscle during prolonged fasting in obese men. Physiol Rep. 2019 Nov;7(21):e14285. doi: 10.14814/phy2.14285. PMID 31724339